CLINICAL TRIAL: NCT07394790
Title: Effectiveness of a Physical Exercise Prescription Program in Primary Care to Improve Physical Fitness and Quality of Life in Adults Aged 65 Years and Older in a Rural Health Area: PREFIS-AP Randomized Controlled Trial
Brief Title: Effectiveness of a Physical Exercise Prescription Program in Primary Care for Adults Aged 65 and Older: PREFIS-AP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREFIS-AP
Record Dates: First submitted 2025-12-12; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Sedentary Lifestyle
Keywords: aging; sarcopenia; Reduced physical fitness
MeSH Terms: conditions — Sedentary Behavior; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned (1:1) to either an individualized exercise prescription program or standard lifestyle advice. Assessors and data analysts will remain blinded to group allocation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Exercise Prescription Program (Experimental): Participants undergo a structured, individualized 12-week Physical Exercise Prescription Program developed after a comprehensive baseline assessment of physical fitness, muscle strength, muscle mass, and physical activity levels. The prescription is generated through the MEDORA Primary Care electronic system and includes five exercise components.
  Interventions: Behavioral: Physical Exercise Prescription Program
- Standard Health Advice (No Intervention): Participants receive general advice to engage in brisk walking on flat terrain for at least 30 minutes daily, consistent with typical Primary Care counseling. No structured exercise plan is provided.

INTERVENTIONS:
Behavioral: Physical Exercise Prescription Program — Participants receive a structured and individualized 12-week program including:
  Aerobic exercise (continuous and interval training, intensity guided by Borg scale)
  Strength training using elastic bands (progressively increasing repetitions, series, and load)
  Respiratory exercises with pressure-based devices
  Flexibility exercises (static stretching routines)
  Balance training (single-leg stance, heel-toe walking, eyes-closed tasks)
  The program is generated through the MEDORA electronic system after baseline evaluation. A certified Exercise Technician provides instruction, supervision, and progression adjustments.
  Arms: Physical Exercise Prescription Program

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of an individualized Physical Exercise Prescription Program delivered in Primary Care for adults aged 65 years and older. The intervention includes a structured assessment of physical fitness, muscle function and mass, physical activity level, and quality of life, followed by a tailored exercise plan encompassing aerobic, strength, respiratory, flexibility, and balance training. Outcomes will be compared with a control group receiving standard health advice to walk briskly for at least 30 minutes daily. The study also explores associations between polypharmacy, muscle function, physical performance, and quality of life.

DETAILED DESCRIPTION:
Sedentary behavior is strongly associated with multiple adverse health outcomes, particularly in older adults. Conventional lifestyle advice alone has shown limited effectiveness in increasing physical activity levels. Exercise prescription delivered through structured evaluation, individualized planning, and scheduled follow-up may lead to clinically significant improvements in physical function and quality of life.

This study will recruit 210 adults aged ≥65 years from a rural Primary Care center. Participants will undergo baseline assessments including sociodemographic variables, anthropometric measures, muscle strength (handgrip dynamometry and chair stand test), aerobic capacity (6-minute walk test), muscle mass (calf circumference and ultrasound of rectus femoris), physical activity level (GPAQ), and quality of life (SF-36). After randomization (1:1), the intervention group will receive a personalized exercise prescription generated through the MEDORA Primary Care electronic system and supervised by a qualified Exercise Technician. The control group will receive routine health advice.

After three months, all participants will be reassessed using the same measures. The study will analyze the effect of the intervention on physical fitness, physical activity, muscle mass and function, and quality of life, including sex-specific differences and the role of polypharmacy. The project incorporates a partial masking strategy and uses REDCap for data management and anonymization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Motivated to participate and able to provide informed consent
* Able to attend baseline assessment and follow-up
* Clinical stability allowing participation in exercise evaluation

Exclusion Criteria:

* Recent myocardial infarction
* Unstable angina
* Uncontrolled arrhythmias (symptomatic or hemodynamically compromising)
* Syncope
* Acute endocarditis, myocarditis, or pericarditis
* Severe or symptomatic aortic stenosis
* Uncontrolled heart failure
* Recent pulmonary thromboembolism or pulmonary infarction
* Lower-limb thrombosis
* Severe aortic stenosis or suspected dissecting aortic aneurysm
* Uncontrolled asthma
* Pulmonary edema
* Acute respiratory failure
* Acute non-cardiopulmonary illness that impairs exercise capacity (e.g., infection, thyrotoxicosis, acute renal failure)
* Mental disorder that prevents adequate cooperation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline to 3 months.
  Quality of Life will be measured by the SF-36 questionnaire. The SF-36 questionnaire is a widely used, patient-reported questionnaire measuring health-related quality of life. It uses points to assess health, with responses on Likert scales (e.g., 0 to 100) transformed into scores for 8 health domains: physical functioning, role limitations (physical/emotional), bodily pain, general health, vitality, social functioning, and mental health, where higher scores mean better health, ranging from 0 (maximum disability) to 100 (no disability).

SECONDARY OUTCOMES:
Physical Activity Level (GPAQ) | Baseline to 3 months.
  Change in physical activity level as measured by the Global Physical Activity Questionnaire (GPAQ), including time spent in work-related activity, transport-related activity, leisure-time activity, and sedentary behavior. Participants will be classified into WHO categories (high, moderate, or low/inactive) based on standardized scoring procedures.
Aerobic Capacity (6-Minute Walk Test) | Baseline to 3 months.
  Change in functional aerobic capacity assessed by the 6-minute walk test (6MWT). The primary variable will be the total distance walked in meters during 6 minutes. Physiological responses (heart rate, oxygen saturation, perceived exertion using Borg scale) will also be recorded.
Muscle Strength - Handgrip Dynamometry | Baseline to 3 months.
  Change in maximal isometric handgrip strength measured with a JAMAR dynamometer (kg), using the highest value from standardized bilateral measurements. Cut-off values will follow European sarcopenia consensus criteria (<27 kg for men; <16 kg for women).
Muscle Strength - Chair Stand Test | Baseline to 3 months.
  Change in lower-limb functional strength measured by the 30-second chair stand test. The outcome is the total number of complete sit-to-stand repetitions performed within 30 seconds following standardized protocol.
Muscle Mass - Calf Circumference | Baseline to 3 months.
  Change in muscle mass estimated by calf circumference (cm), measured at the widest point of the calf using a flexible tape. A value <31 cm will be considered indicative of potential muscle mass deficit.
Muscle Mass - Ultrasound of Rectus Femoris | Baseline to 3 months.
  Change in quantitative and qualitative muscle parameters assessed by ultrasound of the rectus femoris (muscle thickness, cross-sectional area, and echogenicity), following validated measurement criteria for sarcopenia assessment.
Sex Differences in Response to the Exercise Prescription Program (Standardized Change Score) | Baseline to 3 months.
  This outcome will assess whether biological sex modifies the effect of the intervention on functional and health-related outcomes. Sex-specific differences will be evaluated using standardized change scores (z-scores).
  The standardized composite score will be derived from the following previously defined outcome measures:
  Muscle strength (handgrip dynamometry (kg) and the 30-second chair stand test) Aerobic capacity (6-minute walk test) Muscle mass, assessed by calf circumference (cm) and ultrasound measurements of rectus femoris muscle thickness Physical activity level, (Global Physical Activity Questionnaire (GPAQ) Health-related quality of life (SF-36 questionnaire) Each variable will be standardized before aggregation to ensure comparability across different units of measurement. The resulting composite score will be compared between men and women to determine if sex influences the magnitude of response to the exercise prescription program.
Correlation Between Polypharmacy and Change in Handgrip Strength | Baseline to 3 months
  This outcome will assess the correlation between baseline medication burden and change in muscle strength in older adults from baseline to 3 months.
  Medication burden will be defined as the total number of chronic medications taken at baseline (unit: number of medications).
  Muscle strength will be assessed by handgrip strength, measured in kilograms (kg) using a calibrated hand dynamometer. Change in handgrip strength will be calculated as the difference between baseline and 3-month values.
Correlation Between Polypharmacy and Change in Appendicular Skeletal Muscle Mass | Baseline to 3 months
  This outcome will assess the correlation between baseline medication burden and change in muscle mass in older adults from baseline to 3 months.
  Medication burden will be defined as the total number of chronic medications taken at baseline (unit: number of medications).
  Muscle mass will be assessed as appendicular skeletal muscle mass, measured in kilograms (kg) using dual-energy X-ray absorptiometry (DXA). Change in muscle mass will be calculated as the difference between baseline and 3-month values.
Correlation Between Polypharmacy and Change in Physical Performance | Baseline to 3 months
  This outcome will assess the correlation between baseline medication burden and change in physical performance in older adults from baseline to 3 months.
  Medication burden will be defined as the total number of chronic medications taken at baseline (unit: number of medications).
  Physical performance will be assessed using the Short Physical Performance Battery (SPPB), reported as a total score (points on a standardized scale). Change in SPPB score will be calculated as the difference between baseline and 3-month values.
Correlation Between Polypharmacy and Change in Quality of Life | Baseline to 3 months
  This outcome will assess the correlation between baseline medication burden and change in quality of life in older adults from baseline to 3 months.
  Medication burden will be defined as the total number of chronic medications taken at baseline (unit: number of medications).
  Quality of life will be assessed using the EuroQol-5 Dimension (EQ-5D) questionnaire, reported as a standardized index score. Change in EQ-5D score will be calculated as the difference between baseline and 3-month values.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud de Villoria, Villoría, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized datasets and analytic code will be available upon reasonable request, following approval by the Ethics Committee and IBSAL data governance board.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available starting 12 months after publication of primary results and for a minimum of 5 years thereafter.
Access Criteria: Qualified researchers with a methodologically sound proposal, as determined by the study steering committee, will be able to access the data. Requests should be directed to the study PI. A data access agreement will be required.